CLINICAL TRIAL: NCT00360230
Title: A Partially-blind (Observer-blind) Study to Evaluate the Safety and Immunogenicity of 3 Different Vaccination Schedules With 2 GSK Biologicals' Candidate Plasmodium Falciparum Vaccines in Children Aged 5 to 17 Months Living in Ghana
Brief Title: Partially-blind (Observer-blind) Study of Safety and Immunogenicity of Two Malaria Vaccines in Ghanaian Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 106367
Record Dates: First submitted 2006-07-31; First posted 2006-08-04 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Malaria
Keywords: Vaccine; Prophylaxis Plasmodium falciparum malaria; Plasmodium falciparum; Malaria
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (7):
- SB257049 F2 0-1 M Group (Experimental): Healthy infants between 5 and 17 months of age at the time of first vaccination received 2 doses of SB257049 formulation 2 (F2) vaccine according to a 0, 1-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- SB257049 F1 0-1 M Group (Experimental): Healthy infants between 5 and 17 months of age at the time of first vaccination received 2 doses of SB257049 formulation 1 (F1) vaccine according to a 0, 1-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- SB257049 F2 0-1-2 M Group (Experimental): Healthy infants between 5 and 17 months of age at the time of first vaccination received 3 doses of SB257049 formulation 2 (F2) vaccine according to a 0, 1, 2-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- SB257049 F1 0-1-2 M Group (Experimental): Healthy infants between 5 and 17 months of age at the time of first vaccination received 3 doses of SB257049 formulation 1 (F1) vaccine according to a 0, 1, 2-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- SB257049 F2 0-1-7 M Group (Experimental): Healthy infants between 5 and 17 months of age at the time of first vaccination received 3 doses of SB257049 formulation 2 (F2) vaccine according to a 0, 1, 7-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- SB257049 F1 0-1-7 M Group (Active Comparator): Healthy infants between 5 and 17 months of age at the time of first vaccination received 3 doses of SB257049 formulation 1 (F1) vaccine according to a 0, 1, 7-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- Rabipur 0-1-2 M Group (Active Comparator): Healthy infants between 5 and 17 months of age at the time of first vaccination received 3 doses of Rabipur vaccine according to a 0, 1, 2-month schedule administered intramuscularly (IM) in the left deltoid muscle.
  Interventions: Biological: Rabipur

INTERVENTIONS:
Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049 — 2 different formulations are tested. For each formulation, 3 different dosing schedules are tested
  Other Names: RTS; S vaccine
  Arms: SB257049 F1 0-1 M Group; SB257049 F1 0-1-2 M Group; SB257049 F1 0-1-7 M Group; SB257049 F2 0-1 M Group; SB257049 F2 0-1-2 M Group; SB257049 F2 0-1-7 M Group
Biological: Rabipur — 3-dose intramuscular injection.
  Arms: Rabipur 0-1-2 M Group

SUMMARY:
This study will investigate the safety and immunogenicity of 2 candidate malaria vaccines administered according to 3 different vaccination schedules in 5 to 17 months old Ghanaian children. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This study will be conducted in a partially blind fashion: it will be observer-blind as to which vaccine was administered, and open as to the vaccination schedule. One group of children on the 0, 1, 2-schedule will receive a Rabies vaccine as a control. One group on the same schedule will receive the RTS,S/AS02D experimental vaccine as an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child between 5 months and 17 months of age at the time of first vaccination.
* Written or oral, signed or thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Proof that child has received a full 3-dose regimen of licensed Hepatitis B vaccine in infancy.

Exclusion Criteria:

* Acute disease at the time of enrolment.
* Serious acute or chronic illness determined by clinical or physical examination and laboratory screening tests.
* Laboratory screening tests for haemoglobin, total white cell count, platelets, ALT and creatinine out of acceptable limits.
* Planned administration/administration of a vaccine (not in the scope of the study) within 30 days of the first dose of vaccine(s) with the exception of tetanus toxoid or scheduled Yellow fever or Measles vaccine.
* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the first dose of the study vaccine, or planned use during the study period.
* Administration of immunoglobulins, blood transfusions or other blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Simultaneous participation in any other clinical trial;
* Previous participation in any other malaria vaccine trial;
* Any twins
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2006-08-30 (Actual); Primary Completion 2007-08-25 (Actual); Study Completion 2008-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Kumasi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ansong D, Asante KP, Vekemans J, Owusu SK, Owusu R, Brobby NA, Dosoo D, Osei-Akoto A, Osei-Kwakye K, Asafo-Adjei E, Boahen KO, Sylverken J, Adjei G, Sambian D, Apanga S, Kayan K, Janssens MH, Lievens MJ, Olivier AC, Jongert E, Dubois P, Savarese BM, Cohen J, Antwi S, Greenwood BM, Evans JA, Agbenyega T, Moris PJ, Owusu-Agyei S. T cell responses to the RTS,S/AS01(E) and RTS,S/AS02(D) malaria candidate vaccines administered according to different schedules to Ghanaian children. PLoS One. 2011 Apr 27;6(4):e18891. doi: 10.1371/journal.pone.0018891. PMID 21556142
- [Background] Owusu-Agyei S, Ansong D, Asante K, Kwarteng Owusu S, Owusu R, Wireko Brobby NA, Dosoo D, Osei Akoto A, Osei-Kwakye K, Adjei EA, Boahen KO, Sylverken J, Adjei G, Sambian D, Apanga S, Kayan K, Vekemans J, Ofori-Anyinam O, Leach A, Lievens M, Demoitie MA, Dubois MC, Cohen J, Ballou WR, Savarese B, Chandramohan D, Gyapong JO, Milligan P, Antwi S, Agbenyega T, Greenwood B, Evans J. Randomized controlled trial of RTS,S/AS02D and RTS,S/AS01E malaria candidate vaccines given according to different schedules in Ghanaian children. PLoS One. 2009 Oct 2;4(10):e7302. doi: 10.1371/journal.pone.0007302. PMID 19806184
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106367 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106367 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106367 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106367 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106367 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106367 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group | Rabipur 0-1-2 M Group
Started | 90 | 90 | 45 | 90 | 90 | 90 | 45
Completed | 84 | 87 | 42 | 88 | 85 | 86 | 43
Not Completed | 6 | 3 | 3 | 2 | 5 | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Migrated | 4 | 1 | 3 | 1 | 4 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- SB257049 F1 0-1 M Group: Healthy infants between 5 and 17 months of age at the time of first vaccination received received 2 doses of SB257049 formulation 1 (F1) vaccine according to a 0, 1-month schedule administered intramuscularly (IM) in the left deltoid muscle.
- Total: Total of all reporting groups
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group | Total
Number analyzed (Participants) | 90 | 90 | 45 | 90 | 45 | 90 | 90 | 540
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.5 (3.4) | 10.4 (3.4) | 11.2 (3.3) | 10.9 (3.7) | 10.9 (3.5) | 10.4 (3.6) | 10.7 (3.3) | 10.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 23 | 40 | 27 | 44 | 48 | 265
  Male | 49 | 48 | 22 | 50 | 18 | 46 | 42 | 275
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 to Month 10
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data are available.
Measure: Count of Participants; unit: Participants
Groups:
- SB257049 F2 0-1 M Group: Healthy infants between 5 and 17 months of age at the time of first vaccination received received 2 doses of SB257049 formulation 2 (F2) vaccine according to a 0, 1-month schedule administered intramuscularly (IM) in the left deltoid muscle.
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
Number analyzed (Participants) | 90 | 90 | 45 | 90 | 45 | 90 | 90
Participants | 10 | 19 | 5 | 13 | 6 | 17 | 14

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 swelling = swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0 - 6) post-vaccination period following each dose and across doses
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data are available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
Number analyzed (Participants) | 90 | 90 | 45 | 90 | 45 | 90 | 90
Participants
  Any Pain, Dose 1 | 61 | 24 | 23 | 23 | 14 | 53 | 38
  Grade 3 Pain, Dose 1 | 8 | 0 | 3 | 1 | 0 | 8 | 1
  Any Swelling, Dose 1 | 26 | 14 | 12 | 6 | 2 | 16 | 15
  Grade 3 Swelling, Dose 1 | 2 | 0 | 0 | 0 | 0 | 5 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Any Pain, Dose 2 | 37 | 28 | 19 | 30 | 10 | 47 | 38
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Grade 3 Pain, Dose 2 | 2 | 0 | 0 | 1 | 0 | 1 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Any Swelling, Dose 2 | 18 | 7 | 11 | 7 | 1 | 16 | 11
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 2 | 0 | 5 | 1
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Any Pain, Dose 3 |  |  | 16 | 27 | 3 | 42 | 40
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Grade 3 Pain, Dose 3 |  |  | 1 | 0 | 0 | 1 | 1
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Any Swelling, Dose 3 |  |  | 24 | 21 | 0 | 17 | 11
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Grade 3 Swelling, Dose 3 |  |  | 1 | 0 | 0 | 3 | 0
  Any Pain, Across Doses | 68 | 41 | 32 | 50 | 21 | 78 | 67
  Grade 3 Pain, Across Doses | 10 | 0 | 4 | 2 | 0 | 9 | 2
  Any Swelling, Across Doses | 35 | 17 | 31 | 28 | 3 | 34 | 25
  Grade 3 Swelling, Across Doses | 2 | 0 | 1 | 2 | 0 | 8 | 2

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0 - 6) post-vaccination period following each dose and across doses
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
Number analyzed (Participants) | 90 | 90 | 45 | 90 | 45 | 90 | 90
Participants
  Any Drowsiness, Dose 1 | 19 | 14 | 13 | 14 | 3 | 21 | 10
  Grade 3 Drowsiness, Dose 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 1 | 18 | 9 | 12 | 11 | 3 | 16 | 7
  Any Fever, Dose 1 | 33 | 24 | 13 | 19 | 5 | 36 | 26
  Grade 3 Fever, Dose 1 | 3 | 3 | 0 | 0 | 1 | 6 | 1
  Related Fever, Dose 1 | 26 | 16 | 12 | 16 | 2 | 27 | 15
  Any Irritability, Dose 1 | 43 | 20 | 17 | 23 | 11 | 50 | 23
  Grade 3 Irritability, Dose 1 | 1 | 2 | 1 | 1 | 0 | 2 | 1
  Related Irritability, Dose 1 | 40 | 14 | 17 | 18 | 9 | 43 | 18
  Any Loss of appetite, Dose 1 | 21 | 16 | 15 | 15 | 9 | 28 | 18
  Grade 3 Loss of appetite, Dose 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1
  Related Loss of appetite, Dose 1 | 14 | 8 | 11 | 11 | 3 | 17 | 11
  Any Drowsiness, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Any Drowsiness, Dose 2 | 7 | 12 | 6 | 12 | 3 | 16 | 13
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Grade 3 Drowsiness, Dose 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Related Drowsiness, Dose 2 | 6 | 10 | 6 | 9 | 2 | 10 | 10
  Any Fever, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Any Fever, Dose 2 | 38 | 39 | 20 | 47 | 8 | 44 | 46
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Grade 3 Fever, Dose 2 | 2 | 2 | 1 | 1 | 1 | 5 | 3
  Related Fever, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Related Fever, Dose 2 | 35 | 37 | 20 | 42 | 3 | 39 | 41
  Any Irritability, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Any Irritability, Dose 2 | 16 | 17 | 9 | 25 | 5 | 28 | 22
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Grade 3 Irritability, Dose 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Related Irritability, Dose 2 | 14 | 15 | 9 | 22 | 2 | 21 | 16
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Any Loss of appetite, Dose 2 | 6 | 12 | 5 | 16 | 4 | 18 | 18
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 90 | 88 | 44 | 90 | 45 | 89 | 88
  Related Loss of appetite, Dose 2 | 5 | 11 | 5 | 12 | 1 | 10 | 14
  Any Drowsiness, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Any Drowsiness, Dose 3 |  |  | 3 | 9 | 1 | 9 | 16
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Grade 3 Drowsiness, Dose 3 |  |  | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Related Drowsiness, Dose 3 |  |  | 3 | 7 | 1 | 8 | 16
  Any Fever, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Any Fever, Dose 3 |  |  | 19 | 31 | 2 | 48 | 51
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Grade 3 Fever, Dose 3 |  |  | 0 | 4 | 0 | 4 | 3
  Related Fever, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Related Fever, Dose 3 |  |  | 19 | 26 | 2 | 46 | 50
  Any Irritability, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Any Irritability, Dose 3 |  |  | 9 | 23 | 1 | 21 | 25
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Grade 3 Irritability, Dose 3 |  |  | 0 | 0 | 0 | 0 | 0
  Related Irritability, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Related Irritability, Dose 3 |  |  | 9 | 17 | 0 | 19 | 25
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Any Loss of appetite, Dose 3 |  |  | 5 | 12 | 1 | 9 | 16
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Grade 3 Loss of appetite, Dose 3 |  |  | 0 | 0 | 0 | 1 | 1
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 0 | 0 | 44 | 90 | 44 | 88 | 85
  Related Loss of appetite, Dose 3 |  |  | 5 | 5 | 1 | 8 | 14
  Any Drowsiness, Across Doses | 23 | 23 | 17 | 23 | 6 | 35 | 33
  Grade 3 Drowsiness, Across Doses | 0 | 1 | 1 | 0 | 0 | 1 | 0
  Related Drowsiness, Across Doses | 22 | 16 | 16 | 17 | 5 | 27 | 29
  Any Fever, Across Doses | 51 | 47 | 33 | 63 | 14 | 69 | 73
  Grade 3 Fever, Across Doses | 5 | 5 | 1 | 5 | 2 | 13 | 7
  Related Fever, Across Doses | 44 | 44 | 33 | 56 | 7 | 67 | 64
  Any Irritability, Across Doses | 49 | 32 | 23 | 47 | 16 | 63 | 45
  Grade 3 Irritability, Across Doses | 2 | 2 | 1 | 1 | 0 | 4 | 1
  Related Irritability, Across Doses | 45 | 26 | 23 | 39 | 11 | 57 | 39
  Any Loss of appetite, Across Doses | 26 | 25 | 18 | 34 | 13 | 42 | 39
  Grade 3 Loss of appetite, Across Doses | 1 | 1 | 0 | 2 | 0 | 2 | 3
  Related Loss of appetite, Across Doses | 19 | 17 | 15 | 21 | 5 | 28 | 32

4. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day (Days 0 - 29) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
Number analyzed (Participants) | 90 | 90 | 45 | 90 | 45 | 90 | 90
Participants | 78 | 82 | 40 | 80 | 41 | 84 | 85

5. Secondary Outcome: Titers for Anti-Circumsporozoite Protein of Plasmodium Falciparum (Anti-CS)
Description: Titers are presented as geometric mean titers (GMTs) and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Day 0, at Month 2, at Month 7 and at Month 10
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
Number analyzed (Participants) | 87 | 86 | 44 | 86 | 43 | 88 | 88
EL.U/mL
  Day 0 | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.4] | 0.3 [0.2 to 0.3] | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.4]
  Month 2: number analyzed (Participants) | 87 | 85 | 43 | 85 | 43 | 87 | 84
  Month 2 | 318.4 [269.1 to 376.8] | 483.4 [395.4 to 590.9] | 366.9 [293.2 to 459.2] | 631.8 [554.3 to 720.2] | 0.4 [0.3 to 0.6] | 25.9 [19.7 to 34.1] | 51.0 [40.4 to 64.4]
  Month 7: number analyzed (Participants) | 85 | 82 | 43 | 86 | 43 | 81 | 83
  Month 7 | 34.5 [26.1 to 45.5] | 52.7 [40.7 to 68.2] | 78.2 [57.9 to 105.6] | 162.3 [134.2 to 196.3] | 0.3 [0.3 to 0.4] | 272.1 [218.5 to 338.8] | 373.0 [311.1 to 447.2]
  Month 10: number analyzed (Participants) | 84 | 84 | 42 | 84 | 43 | 83 | 84
  Month 10 | 19.9 [14.8 to 26.8] | 30.5 [23.2 to 40.1] | 43.4 [31.6 to 59.6] | 102.1 [83.4 to 125.1] | 0.3 [0.3 to 0.4] | 120.0 [92.2 to 156.1] | 166.5 [140.1 to 198.0]

6. Secondary Outcome: Titers for Anti-Hepatitis B (Anti-HBs)
Description: Titers are presented as geometric mean titers (GMTs) and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Day 0 and at Month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
Number analyzed (Participants) | 87 | 86 | 44 | 86 | 43 | 88 | 88
mIU/mL
  Day 0 | 100.8 [68.3 to 148.8] | 107.6 [73.5 to 157.6] | 108.7 [60.6 to 194.8] | 82.1 [61.0 to 110.5] | 107.9 [63.5 to 183.3] | 88.1 [60.7 to 128.0] | 89.9 [60.8 to 132.7]
  Month 2: number analyzed (Participants) | 87 | 85 | 43 | 85 | 43 | 81 | 83
  Month 2 | 17042.9 [10466.7 to 27750.8] | 15106.5 [9508.4 to 24000.6] | 29999.7 [18798.9 to 47874.2] | 34935.1 [25177.9 to 48473.6] | 121.7 [63.2 to 234.5] | 96754.4 [72062.0 to 129907.7] | 103224.8 [83034.7 to 128324.1]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day post-vaccination period (Days 0-6); Unsolicited AEs: during the 30-day post-vaccination period (Days 0-29); SAEs: during the entire study period (Day 0 - Month 19).
Arm/Group | SB257049 F2 0-1 M Group | SB257049 F1 0-1 M Group | SB257049 F2 0-1-2 M Group | SB257049 F1 0-1-2 M Group | Rabipur 0-1-2 M Group | SB257049 F2 0-1-7 M Group | SB257049 F1 0-1-7 M Group
All-Cause Mortality (participants affected / at risk) | 0/90 | 1/90 | 0/45 | 0/90 | 1/45 | 0/90 | 2/90
Serious Adverse Events (participants affected / at risk) | 18/90 | 23/90 | 11/45 | 22/90 | 7/45 | 24/90 | 17/90
Other Adverse Events (participants affected / at risk) | 85/90 | 87/90 | 44/45 | 89/90 | 43/45 | 89/90 | 89/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB257049 F2 0-1 M Group (N=90) | SB257049 F1 0-1 M Group (N=90) | SB257049 F2 0-1-2 M Group (N=45) | SB257049 F1 0-1-2 M Group (N=90) | Rabipur 0-1-2 M Group (N=45) | SB257049 F2 0-1-7 M Group (N=90) | SB257049 F1 0-1-7 M Group (N=90)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 9 (9) | 1 (1) | 4 (4) | 3 (3) | 9 (9) | 5 (5)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cerebral malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 10 (10) | 0 (0) | 3 (3) | 5 (5)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 9 (9) | 6 (7) | 5 (5) | 6 (7) | 4 (5) | 6 (6) | 6 (6)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 4 (4) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 6 (7) | 4 (6) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 3 (4)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB257049 F2 0-1 M Group (N=90) | SB257049 F1 0-1 M Group (N=90) | SB257049 F2 0-1-2 M Group (N=45) | SB257049 F1 0-1-2 M Group (N=90) | Rabipur 0-1-2 M Group (N=45) | SB257049 F2 0-1-7 M Group (N=90) | SB257049 F1 0-1-7 M Group (N=90)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 3 (3) | 8 (8) | 6 (7) | 3 (3) | 5 (5)
Bronchopneumonia (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 6 (6) | 10 (10) | 3 (3) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 26 (27) | 25 (28) | 18 (25) | 34 (43) | 13 (14) | 42 (55) | 39 (52)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (7) | 0 (0) | 5 (6) | 5 (5) | 8 (10) | 9 (10)
Dysentery (Infections and infestations) | 3 (3) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Eating disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Gastroenteritis (Infections and infestations) | 19 (19) | 27 (27) | 13 (14) | 28 (31) | 9 (9) | 28 (33) | 23 (27)
Impetigo (Infections and infestations) | 7 (7) | 2 (2) | 0 (0) | 11 (12) | 5 (5) | 15 (16) | 12 (13)
Irritability (Psychiatric disorders) | 49 (59) | 32 (37) | 23 (35) | 47 (71) | 16 (17) | 63 (99) | 45 (70)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 6 (6)
Malaria (Infections and infestations) | 24 (29) | 23 (26) | 15 (16) | 24 (25) | 17 (17) | 30 (32) | 27 (31)
Otitis media (Infections and infestations) | 2 (2) | 2 (2) | 4 (5) | 5 (6) | 1 (1) | 8 (9) | 10 (10)
Pain (General disorders) | 68 (98) | 41 (52) | 32 (58) | 50 (80) | 21 (27) | 78 (142) | 67 (116)
Plasmodium falciparum infection (Infections and infestations) | 12 (12) | 8 (8) | 2 (2) | 11 (11) | 13 (15) | 14 (16) | 15 (17)
Pyrexia (General disorders) | 52 (72) | 47 (63) | 33 (52) | 63 (98) | 14 (15) | 69 (128) | 73 (123)
Respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 3 (3) | 8 (8) | 2 (2) | 7 (9) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 6 (6) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 23 (26) | 23 (26) | 17 (22) | 23 (35) | 6 (7) | 35 (46) | 33 (39)
Swelling (General disorders) | 35 (44) | 17 (21) | 31 (47) | 28 (34) | 3 (3) | 34 (49) | 25 (37)
Upper respiratory tract infection (Infections and infestations) | 39 (46) | 49 (60) | 28 (36) | 45 (64) | 25 (38) | 49 (62) | 49 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.